CLINICAL TRIAL: NCT01966302
Title: Compassionate Use of Beraprost Sodium 314d Modified Release (BPS-314d-MR) for Three Patients With Pulmonary Arterial Hypertension (PAH).
Brief Title: Compassionate Use of Beraprost Sodium 314d Modified Release for Patients With Pulmonary Arterial Hypertension (PAH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Collaborators: Lung Biotechnology PBC (Industry)
Responsible Party: Principal Investigator, ronald oudiz, m.d., Professor of Medicine, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Compassionate use BPS-314d-MR
Record Dates: First submitted 2013-10-15; First posted 2013-10-21 (Estimated); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension; prostacyclin; oral
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — beraprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Beraprost open label (Experimental): Compassionate use access to open label BPS-314d-MR
  Interventions: Drug: BPS-314d-MR

INTERVENTIONS:
Drug: BPS-314d-MR — 15-150 mcg po BID,
  Other Names: Beraprost 314-d modified release

SUMMARY:
The purpose of this study is to see if Lung LLC's new experimental formulation of the medicine Beraprost Sodium, called Beraprost Sodium 314d Modified Release (BPS-314d-MR), can improve the symptoms of pulmonary arterial hypertension (PAH) in patients. An experimental drug is one that has not been approved by the U.S. Food and Drug Administration for use in the general public. This research study is for patients who have pulmonary arterial hypertension (PAH) and have just completed taking part in an earlier research study and received an older experimental formulation of Beraprost Sodium, called Beraprost Sodium Modified Release (BPS-MR). That earlier study was being done to see if BPS-MR could improve their PAH.

Patients may also be taking Tyvaso (treprostinil), Tracleer (bosentan), Letairis (ambrisentan), Adcirca (tadalafil) and/or Viagra or Revatio (sildenafil) to treat their PAH. The diagnosis of PAH means that the blood pressure in their lungs is higher than normal. The increased blood pressure in the lungs places a strain on the heart. The strain causes the heart to pump less blood into the lungs, causing shortness of breath and tiredness. The strain on the heart weakens the heart muscle making it less able to pump blood, a condition called heart failure. As heart failure develops, swelling in the feet and abdomen may occur.

DETAILED DESCRIPTION:
According to Lung LLC, and from my review of summary results contained within the most recent version of the BPS-314d-MR Investigators' Brochure I concur, BPS-314d- MR has been shown to have a similar safety and pharmacokinetic profile in healthy volunteers to BPS-MR. It is also my understanding that at an End of Phase II meeting in April of this year, FDA acknowledged Lung LLC's intention to continue the development of BPS-314d-MR by conducting a Phase III pivotal study in PAH patients. This study, BPS-314d-MR-PAH-302 was subsequently initiated this past June.

In my opinion, and based upon the similarities of the two formulations, it is in the best interest of our patients to transition their treatment to BPS-314d-MR.

Lung LLC has agreed to supply BPS-314d-MR for the patients.

ELIGIBILITY:
Inclusion Criteria:

* Prior participation in Beraprost-MR study at Harbor-UCLA

Exclusion Criteria:

* No prior participation in Beraprost study at Harbor-UCLA

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2019-06-02 (Actual); Study Completion 2019-06-02 (Actual)

PRIMARY OUTCOMES:
Number of participants experiencing Adverse Events | 2 years
  To determine the overall safety of open label study drug by tabulating the number of patients experiencing Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Ronald J Oudiz, MD, Principal Investigator — Los Angeles BRI
Locations (1):
- Los Angeles Biomedical research Institute, Torrance, California, United States